CLINICAL TRIAL: NCT02536313
Title: A Phase 2, Open-Label Study to Investigate the Safety and Efficacy of Sofosbuvir/GS-5816/GS-9857 Fixed-Dose Combination With or Without Ribavirin in Subjects With Chronic Genotype 1 HCV Infection Previously Treated With a Direct Acting Antiviral Regimen
Brief Title: Safety and Efficacy of Sofosbuvir/Velpatasvir/Voxilaprevir Fixed-Dose Combination With or Without Ribavirin in Participants With Chronic Genotype 1 HCV Infection Previously Treated With a Direct Acting Antiviral Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-367-1871
Record Dates: First submitted 2015-08-27; First posted 2015-08-31 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir velpatasvir voxilaprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SOF/VEL/VOX (Experimental): SOF/VEL/VOX for 12 weeks
  Interventions: Drug: SOF/VEL/VOX
- SOF/VEL/VOX + RBV (Experimental): SOF/VEL/VOX + RBV for 12 weeks
  Interventions: Drug: SOF/VEL/VOX; Drug: RBV

INTERVENTIONS:
Drug: SOF/VEL/VOX — 400/100/100 mg FDC tablet administered orally once daily with food
  Other Names: GS-7977/GS-5816/GS-9857; Vosevi®
Drug: RBV — Tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: SOF/VEL/VOX + RBV

SUMMARY:
The primary objective of this study is to evaluate the efficacy, safety, and tolerability of the treatment with sofosbuvir/velpatasvir/voxilaprevir (SOF/VEL/VOX) fixed dose combination (FDC) ± ribavirin (RBV) in participants with chronic genotype 1 hepatitis C virus (HCV) infection and prior treatment experience with a direct acting antiviral (DAA).

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals with chronic HCV genotype 1 infection
* Documented as treatment experienced with a direct acting antiviral-containing regimen without achieving sustained viral response
* Absence of cirrhosis or presence of compensated cirrhosis
* Screening laboratory values within defined thresholds
* Must use specific contraceptive methods if female of childbearing potential or sexually active male

Key Exclusion Criteria:

* Co-infection with HIV or hepatitis B virus (HBV)
* Current or prior history of clinical hepatic decompensation
* Chronic use of systemic immunosuppressive agents
* History of clinically significant illness or any other medical disorder that may interfere with individual's treatment, assessment or compliance with the protocol
* Pregnant or a nursing female

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2016-03-28 (Actual); Study Completion 2016-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- The Texas Liver Institute, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/about/ethics-and-code-of-conduct/policies.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/about/ethics-and-code-of-conduct/policies

REFERENCES:
- [Background] Lawitz E, Poordad F, Wells J, Hyland RH, Yang Y, Dvory-Sobol H, Stamm LM, Brainard DM, McHutchison JG, Landaverde C, Gutierrez J. Sofosbuvir-velpatasvir-voxilaprevir with or without ribavirin in direct-acting antiviral-experienced patients with genotype 1 hepatitis C virus. Hepatology. 2017 Jun;65(6):1803-1809. doi: 10.1002/hep.29130. Epub 2017 May 3. PMID 28220512

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1 study site in the United States. The first participant was screened on 29 July 2015. The last study visit occurred on 28 June 2016.
Groups:
- SOF/VEL/VOX: Sofosbuvir/velpatasvir/voxilaprevir (Vosevi®; SOF/VEL/VOX ) (400/100/100 mg) fixed dose combination (FDC) tablet orally once daily with food for 12 weeks
- SOF/VEL/VOX + RBV: SOF/VEL/VOX (400/100/100 mg) FDC tablet + Ribavirin (RBV) (1000 or 1200 mg daily based on weight) tablet orally once daily with food for 12 weeks
Period: Overall Study
Arm/Group | SOF/VEL/VOX | SOF/VEL/VOX + RBV
Started | 24 | 25
Completed | 24 | 24
Not Completed | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who took at least 1 dose of study drug
Groups:
- SOF/VEL/VOX: SOF/VEL/VOX (400/100/100 mg) FDC tablet orally once daily with food for 12 weeks
- SOF/VEL/VOX + RBV: SOF/VEL/VOX (400/100/100 mg) FDC tablet + RBV (1000 or 1200 mg daily based on weight) tablet orally once daily with food for 12 weeks
- Total: Total of all reporting groups
Arm/Group | SOF/VEL/VOX | SOF/VEL/VOX + RBV | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10.1) | 54 (14.1) | 54 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 16 | 16 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 7 | 3 | 10
  White | 17 | 22 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 16 | 17 | 33
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 2 | 5 | 7
    CT | 10 | 13 | 23
    TT | 12 | 7 | 19
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.2 (0.42) | 6.3 (0.46) | 6.3 (0.44)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 4 | 5 | 9
  ≥ 800,000 IU/mL | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Cessation of Treatment (SVR12)
Description: SVR12 is defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: all randomized/enrolled participants who took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | SOF/VEL/VOX | SOF/VEL/VOX + RBV
Number analyzed (Participants) | 24 | 25
percentage of particpants | 100.0 [85.8 to 100.0] | 96.0 [79.6 to 99.9]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued SOF/VEL/VOX Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set: participants who took at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX | SOF/VEL/VOX + RBV
Number analyzed (Participants) | 24 | 25
percentage of participants | 0 | 0

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 are defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOF/VEL/VOX: SOF/VEL/VOX (400/100/100 mg) FDC tablet once daily with food for 12 weeks
- SOF/VEL/VOX + RBV: SOF/VEL/VOX (400/100/100 mg) FDC tablet + RBV (1000 or 1200 mg daily based on weight) tablet once daily with food for 12 weeks
Arm/Group | SOF/VEL/VOX | SOF/VEL/VOX + RBV
Number analyzed (Participants) | 24 | 25
percentage of participants
  SVR4 | 100.0 [85.8 to 100.0] | 96.0 [79.6 to 99.9]
  SVR24 | 100.0 [85.8 to 100.0] | 96.0 [79.6 to 99.9]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment
Time Frame: Weeks 1, 2, 4, 8 and 12
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX | SOF/VEL/VOX + RBV
Number analyzed (Participants) | 24 | 25
percentage of participants
  Week 1 | 54.2 [32.8 to 74.4] | 40 [21.1 to 61.3]
  Week 2 | 79.2 [57.8 to 92.9] | 60.0 [38.7 to 78.9]
  Week 4 | 100 [85.8 to 100.0] | 92.0 [74.0 to 99.0]
  Week 8 | 100.0 [85.8 to 100.0] | 100.0 [86.3 to 100.0]
  Week 12 | 100.0 [85.8 to 100.0] | 100.0 [86.3 to 100.0]

5. Secondary Outcome: HCV RNA Change From Baseline/Day 1 Through Week 12
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL/VOX | SOF/VEL/VOX + RBV
Number analyzed (Participants) | 24 | 25
log10 IU/mL
  Change at Week 1: number analyzed (Participants) | 24 | 24
  Change at Week 1 | -4.63 (0.737) | -4.53 (0.687)
  Change at Week 2 | -4.97 (0.484) | -4.95 (0.566)
  Change at Week 4 | -5.10 (0.419) | -5.14 (0.477)
  Change at Week 8 | -5.10 (0.419) | -5.18 (0.461)
  Change at Week 12 | -5.10 (0.419) | -5.18 (0.461)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure is defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX | SOF/VEL/VOX + RBV
Number analyzed (Participants) | 24 | 25
percentage of participants | 0 | 4.0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks + 30 days
Description: Safety Analysis Set: participants who took at least 1 dose of study drug
Groups:
- SOF/VEL/VOX: SOF/VEL/VOX (400/100/100 mg) tablet orally once daily for 12 weeks
- SOF/VEL/VOX + RBV: SOF/VEL/VOX (400/100/100 mg) tablet + RBV (1000 or 1200 mg daily based on weight) tablet orally once daily for 12 weeks
Arm/Group | SOF/VEL/VOX | SOF/VEL/VOX + RBV
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/25
Other Adverse Events (participants affected / at risk) | 6/24 | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL/VOX (N=24) | SOF/VEL/VOX + RBV (N=25)
Pneumonia (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL/VOX (N=24) | SOF/VEL/VOX + RBV (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 0 | 9
Bronchitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years